CLINICAL TRIAL: NCT06864195
Title: Development of a Breath Test Using Volatile Organic Markers for Monitoring Cirrhosis and Detecting Primary Liver Tumours (VOCAL2)
Brief Title: A Simple Breath Test to Detect Liver Cancer and Monitor Liver Conditions
Acronym: VOCAL2
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 175288
Record Dates: First submitted 2025-02-20; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Liver Cirrhosis; Hepatocellular Carcinoma (HCC); Cholangiocarcinoma; Cholangitis, Sclerosing
Keywords: breath; liver cancer; cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Cholangiocarcinoma; Cholangitis, Sclerosing; Liver Neoplasms; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- participants with liver cancer: Histologically or radiologically-confirmed hepatocellular carcinoma or cholangiocarcinoma
- participants with benign liver disorders: 1. Liver cirrhosis, confirmed on imaging or histology from biopsy or
  2. Primary sclerosing cholangitis, confirmed on MRCP/ERCP or histology from biopsy
- healthy controls: Non-specific gastrointestinal symptoms, but a radiologically-normal liver

SUMMARY:
Liver cancer is often diagnosed too late for effective treatment. The VOCAL2 study is developing a simple, non-invasive breath test to help detect liver cancer earlier and monitor liver conditions like cirrhosis. The test analyzes tiny chemicals in exhaled breath called volatile organic compounds (VOCs) to identify signs of liver disease.

Who can take part?

Adults aged 18 or older who:

Have liver cancer (hepatocellular carcinoma or cholangiocarcinoma), or Have liver cirrhosis or primary sclerosing cholangitis, or Have tummy symptoms but a normal liver scan. What's involved?

Participants will:

Give a breath sample after fasting for 6 hours. Answer a few health questions. Allow access to relevant medical records. The appointment lasts about 1 hour at an NHS hospital. Benefits & Risks

This research could lead to an earlier, easier way to detect liver cancer, but there's no direct health benefit for participants.

There are no risks, as breath sampling is completely non-invasive and safe. Where is the study happening? Led by Imperial College London, running in NHS hospitals across the UK.

Who is funding the study? The study is funded by Rosetrees and Stoneygate Trust.

Contact Information Email: vocal-study@imperial.ac.uk Phone: +44 (0)20 7594 3396

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Adult participants ≥ 18 years old
* Participants with either:

  1. Histologically or radiologically-confirmed* hepatocellular carcinoma or cholangiocarcinoma (participants with liver cancer)
  2. Liver cirrhosis, confirmed on imaging or histology from biopsy (participants with benign liver disorders)
  3. Primary sclerosing cholangitis, confirmed on MRCP/ERCP or histology from biopsy (participants with benign liver disorders)
  4. Non-specific gastrointestinal symptoms, but a radiologically-normal liver (healthy controls)

Exclusion Criteria:

* Active infection, or receiving immunosuppressive medications, within the preceding eight weeks
* History of another cancer within the previous five years
* Previous liver resection
* Already received chemotherapy, radiotherapy or surgery for their liver cancer
* Comorbidities preventing breath collection
* Pregnant women (checked verbally with participant).
* Unable to provide informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People from secondary or tertiary centers
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of VOC Analysis for Liver Cancer Detection | Day 1
  This outcome measures the ability of volatile organic compound (VOC) analysis in exhaled breath to accurately detect liver cancer. Breath samples will be analysed using thermal desorption gas chromatography-mass spectrometry (TD-GC-MS). The diagnostic accuracy will be determined by comparing VOC profiles with histological confirmation or radiological imaging as the reference standard. Sensitivity, specificity, and area under the receiver operating characteristic curve (AU-ROC) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: George Hanna, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.wcrf.org/cancer-trends/liver-cancer-statistics/
- See also: Related Info — https://www.cancerresearchuk.org/health-professional/cancer-statistics/statistics-by-cancer-type/liver-cancer